CLINICAL TRIAL: NCT04013776
Title: The Impact of a Low or High Phosphate Diet on Phosphate and Calcium Excretion in Healthy People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Rachel Holden, Professor of Medicine Queen's University, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DMED-2031-17
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; Aging; Nutrient; Excess
MeSH Terms: conditions — Cardiovascular Diseases | interventions — sodium phosphate

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phosphate supplemented diet (Active Comparator): All participants will undergo phosphate testing after following a phosphate supplemented diet for 5 days
  Interventions: Dietary Supplement: Phosphate supplemented diet
- Low phosphate diet (No Intervention): All participants will undergo phosphate testing after following a low phosphate diet for 5 days

INTERVENTIONS:
Dietary Supplement: Phosphate supplemented diet — Participants will be asked to follow a 5 day menu of 750 mg of phosphorus daily along with a daily sodium phosphorus supplement of 500 mg
  Other Names: sodium phosphate
  Arms: Phosphate supplemented diet

SUMMARY:
Phosphate is present in many of the foods that the investigators eat and is required by many cellular processes. The kidneys are the only organ that excrete the extra phosphate from the diet that the body does not require. Phosphate is linked to vascular calcification and cardiovascular disease. Measures of serum phosphate do not reflect the burden of phosphate and are not sensitive to early changes in the way the kidneys eliminate phosphate. This study will determine whether the kidneys handle an oral phosphate load differently after 5 days of a low phosphate diet compared to 5 days of a high phosphate diet.

DETAILED DESCRIPTION:
In this study, participants will follow a low-phosphorus diet (750 mg) with a 500 mg calcium supplement for 5 days keeping a detailed diary of the foods eaten during this period. On the 5th day, the participant will undergo a 24 hour urine collection. Participants will present after an overnight fast for baseline blood and urine measurements. Then they will consume water containing 500 mg of phosphorus. Urine and blood will be collected every hour for 3 hours for measurement of phosphate and calcium and for measurement of hormones known to regulate phosphate and calcium including fibroblast growth factor-23, parathyroid hormone and vitamin D. One week later, participants will follow the same diet but will also receive a 1250 mg phosphorus supplement for 5 days. On the 5th day, urine will be collected for 24 hours. Participants will present again after an overnight fast and undergo the identical testing.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* between ages of 20 and 40

Exclusion Criteria:

* known heart disease
* known diabetes
* pregnant
* breast-feeding

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Urinary phosphate excretion | 3 hours
  Change in urinary phosphate excretion after 500 mg phosphorus challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No